CLINICAL TRIAL: NCT01370304
Title: Repetitive Transcranial Magnetic Stimulation (rTMS) Compared or Associated With Venlafaxine for Depressive Disorder: A Functional Magnetic Resonance Imaging (fMRI) Study
Brief Title: Repetitive Transcranial Magnetic Stimulation Compared or Associated With Venlafaxine for Depressive Disorder
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Principal Investigator, fengshufang, Fourth Military Medical University, Department of Psychosomatics, Xijing Hospital, Xijing Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20110526-09
Record Dates: First submitted 2011-06-08; First posted 2011-06-09 (Estimated); Last update posted 2012-02-15 (Estimated); Status verified 2012-02

CONDITIONS: Depression
Keywords: repetitive Transcranial Magnetic Stimulation (rTMS); Depression; Venlafaxine; fMRI
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- active rTMS and active Venlafaxine (Experimental)
  Interventions: Other: active rTMS and active Venlafaxine
- active rTMS and sham Venlafaxine (Experimental)
  Interventions: Other: active rTMS and sham Venlafaxine
- sham rTMS and active Venlafaxine (Sham Comparator)
  Interventions: Other: sham rTMS and active Venlafaxine

INTERVENTIONS:
Other: active rTMS and active Venlafaxine — rTMS parameters : Intensity of 120% of individually determined motor threshold; frequency : 1 Hz; 360 impulsions; on period : 1 min; off period : 30 s.5 sessions per week for 4-6 weeks
  Venlafaxine: LP:75mg:1capsule per day for 3 days, then 2 per day for 2 to 4 weeks, if necessary 3 per day the next 2 weeks
  Other Names: venlafaxine: Wyeth; rTMS: MagVenture
  Arms: active rTMS and active Venlafaxine
Other: active rTMS and sham Venlafaxine — rTMS parameters : Intensity of 120% of individually determined motor threshold; frequency : 1 Hz; 360 impulsions; on period : 1 min; off period : 30 s. 5 sessions per week for 4-6 weeks
  Other Names: venlafaxine: Wyeth; rTMS: MagVenture
  Arms: active rTMS and sham Venlafaxine
Other: sham rTMS and active Venlafaxine — rTMS parameters :same coil, same number of pulses but using an angled coil(90 degree)over the frontotemporal region
  Venlafaxine: LP:75mg:1capsule per day for 3 days, then 2 per day for 2 to 4 weeks, if necessary 3 per day the next 2 weeks
  Other Names: venlafaxine: Wyeth; rTMS: MagVenture
  Arms: sham rTMS and active Venlafaxine

SUMMARY:
The purpose of this study is to treat participants with a diagnosis of depressive disorder to assess the efficacy of repetitive Transcranial Magnetic Stimulation (rTMS) and venlafaxine in the treatment of depressive disorders compared venlafaxine only (the optimal medication) and to rTMS only. fMRI will be performed to determine if treatment response is related to changes in fMRI, and use it to investigate the respondence to the treatments.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* Clinical diagnosis of major depressive disorder (DSM-IV)
* HDRS-17 items > 20
* Failure of one antidepressant treatment (efficacious doses for 6 weeks at least)

Exclusion Criteria:

* Psychotic features
* Failure of one previous venlafaxine treatment
* Addiction comorbidity or schizophrenia comorbidity
* Involuntary hospitalization
* Seizures history
* Pregnancy or breastfeeding
* Somatic comorbidity able to impact on cognitive functions

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2011-06; Primary Completion 2012-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
The primary outcome measure is remission | 1-6 weeks
  It will be evaluated using the Hamilton Depression Rating Scale (HDRS-17 < 8)

SECONDARY OUTCOMES:
fMRI | 0,6 weeks
CGI | 1-6 weeks
  Using the Clinical Global Impression scale(CGI)
QIDS-C30 | 1-6 weeks
UKU Scale | 1-6 weeks
  Side effects will be assessed using the UKU Scale

CONTACTS AND LOCATIONS:
Overall Officials: Qingrong Tan, Ph.D, Study Chair — Department of Psychiatry, Xi Jing hospital, Xi'an, China
Locations (1):
- Yun chun Chen, Xi'an, Shaanxi, China